CLINICAL TRIAL: NCT03668262
Title: ED50 of Cis-atracurium for Laryngeal Mask Incubation in General Anesthesia During Urology Surgery
Brief Title: ED50 of Cis-atracurium for Laryngeal Mask Incubation in General Anesthesia
Status: Completed | Type: Observational
Sponsor: China International Neuroscience Institution (Other)
Responsible Party: Sponsor
Other Study IDs: CINI-AD-20180808
Record Dates: First submitted 2018-09-11; First posted 2018-09-12 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Urologic Diseases
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- 0.15mg/ kg group: Administration method of cis-atracurium: the dose of the first patient is 0.15 mg / kg, and the ratio between adjacent doses is 1.5. If the laryngeal mask insertion condition of this patient is satisfactory, the next patient will use the lower dose. If the laryngeal mask insertion condition of this patient is not satisfactory, the next patient will use a higher dose. Starting from the first case of dissatisfaction, the number of observation units is counted. Dissatisfaction - satisfaction occurs at 7 exchange points and then the test ends.
  Interventions: Drug: Cis-atracurium
- 0.1mg/ kg group: Administration method of cis-atracurium: the dose of the first patient is 0.15 mg / kg, and the ratio between adjacent doses is 1.5. 0.15/1.5=0.1 ( If the laryngeal mask insertion condition of this patient is satisfactory, the next patient will use the lower dose. If the laryngeal mask insertion condition of this patient is not satisfactory, the next patient will use a higher dose. Starting from the first case of dissatisfaction, the number of observation units is counted. Dissatisfaction - satisfaction occurs at 7 exchange points and then the test ends.)
  Interventions: Drug: Cis-atracurium
- 0.07mg/ kg group: Administration method of cis-atracurium: the dose of the first patient is 0.15 mg / kg, and the ratio between adjacent doses is 1.5. 0.1/1.5=0.0667 ( If the laryngeal mask insertion condition of this patient is satisfactory, the next patient will use the lower dose. If the laryngeal mask insertion condition of this patient is not satisfactory, the next patient will use a higher dose. Starting from the first case of dissatisfaction, the number of observation units is counted. Dissatisfaction - satisfaction occurs at 7 exchange points and then the test ends.)
  Interventions: Drug: Cis-atracurium
- 0.05mg/ kg group: Administration method of cis-atracurium: the dose of the first patient is 0.15 mg / kg, and the ratio between adjacent doses is 1.5. 0.07/1.5=0.0466( If the laryngeal mask insertion condition of this patient is satisfactory, the next patient will use the lower dose. If the laryngeal mask insertion condition of this patient is not satisfactory, the next patient will use a higher dose. Starting from the first case of dissatisfaction, the number of observation units is counted. Dissatisfaction - satisfaction occurs at 7 exchange points and then the test ends.)
  Interventions: Drug: Cis-atracurium
- 0.03mg/ kg group: Administration method of cis-atracurium: the dose of the first patient is 0.15 mg / kg, and the ratio between adjacent doses is 1.5. 0.05/1.5=0.0333 ( If the laryngeal mask insertion condition of this patient is satisfactory, the next patient will use the lower dose. If the laryngeal mask insertion condition of this patient is not satisfactory, the next patient will use a higher dose. Starting from the first case of dissatisfaction, the number of observation units is counted. Dissatisfaction - satisfaction occurs at 7 exchange points and then the test ends.)
  Interventions: Drug: Cis-atracurium
- 0.02mg/ kg group: Administration method of cis-atracurium: the dose of the first patient is 0.15 mg / kg, and the ratio between adjacent doses is 1.5. 0.03/1.5=0.02( If the laryngeal mask insertion condition of this patient is satisfactory, the next patient will use the lower dose. If the laryngeal mask insertion condition of this patient is not satisfactory, the next patient will use a higher dose. Starting from the first case of dissatisfaction, the number of observation units is counted. Dissatisfaction - satisfaction occurs at 7 exchange points and then the test ends.)
  Interventions: Drug: Cis-atracurium

INTERVENTIONS:
Drug: Cis-atracurium — Different concentration of cis-atracurium
  Other Names: muscle relaxants

SUMMARY:
1. The muscle relaxants can improve the conditions of laryngeal mask incubation and reduce the related complications (such as laryngeal spasm and postoperative throat pain)
2. The dosages of muscle relaxants used in various researches vary greatly.
3. We are planning use the most classical method for determining the ED50 or half effective concentration of cis-atracurium using sequential method, which is also called " up and down method" and " ladder method".

DETAILED DESCRIPTION:
The concordance of the current research is that muscle relaxants can improve the conditions of laryngeal mask incubation and reduce the related complications (such as laryngeal spasm and postoperative throat pain ) of laryngeal mask incubation. It is necessary to use muscle relaxants in laryngeal mask incubation under non-special circumstances. However, the dosages of muscle relaxants used in various researches vary greatly of normal endotracheal intubation. Previous studies have shown that the amount of muscle relaxant required for laryngeal mask intubation is smaller than that required for endotracheal intubation. Although the dosage of muscle relaxant required for tracheal intubation can ensure the smooth insertion of laryngeal mask airway, laryngeal mask airway is mostly used for short surgery, which is prone to postoperative muscle relaxation residue and prolongs the recovery. We planning use the most classical method for determining the ED50 or half effective concentration of cis-atracurium using sequential method, which is also called " up and down method" and " ladder method".

ELIGIBILITY:
Inclusion Criteria:

1. ASA Ⅱ~Ⅲlevel;
2. BMI18.5-30；
3. Those who intend to undergo short urological surgery ( operation time < 1h );
4. Age 25~75 years
5. Estimated amount of bleeding < 5ml / kg.

Exclusion Criteria:

1. Neuromuscular diseases or metabolic diseases;
2. Preoperative complicated with water and electrolytes disorders ( such as hypokalemia and hypocalcemia );
3. Serious hepatic and renal insufficiency and serious heart and lung diseases;
4. Predictable difficult airway;
5. Take drugs ( such as aminoglycoside, polymyxin, phenytoin sodium, carbamazepine, etc. ) that affect the nerve-muscle transmission function or the efficacy of muscle relaxants before surgery;
6. Muscle relaxation drug allergy;
7. Previous history of alcoholism or drug abuse.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients in Xuanwu Hospital for elective short urological surgery are selected.
  One day before surgery, visitors recorded basic information such as the patient's sex, age, BMI, ASA grade in the ward, carried out airway evaluation, and recorded the mouth opening to make sure they can be included
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Laryngeal mask insertion conditions(satisfactory/unsatisfactory) | through study completion, an average of 1 day
  The evaluation criteria of laryngeal mask insertion conditions are based on siva lingam's six-point three-level table, which is evaluated from the following six aspects: the degree of mouth opening, difficulty in laryngeal mask insertion, cough, retch, laryngeal spasm, and body movement. Each item is divided into 3, 2 and 1 points according to the degree of severity, with a full score of 18 points, 16 points and above being satisfactory, and 16 points and below being unsatisfactory.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang X, Huang K, Yan H, Lan F, Yao D, Li Y, Xue J, Wang T. The median effective dose (ED50) of cis-Atracurium for laryngeal mask airway insertion during general Anaesthesia for patients undergoing urinary surgery. BMC Anesthesiol. 2020 Mar 19;20(1):68. doi: 10.1186/s12871-020-00982-3. PMID 32192431